CLINICAL TRIAL: NCT06242860
Title: A Prospective, Clinical Trial Eye Lipid Mobilizer (ELM) Using Heat and Vibration for the Treatment of Meibomian Gland Dysfunction (MGD)
Brief Title: Clinical Study Using Eye Lipid Mobilizer (ELM) With Heat and Vibration To Treat Evaporative Dry Eye Disease
Acronym: ELM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eyedetec Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTL 1011
Record Dates: First submitted 2024-01-19; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Evaporative Dry Eye Disease; Meibomian Gland Dysfunction
Keywords: dry eye disease; meibomian gland dysfunction; evaporative dry eye disease; eye lipid mobilizer
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Single ELM Treatment (Active Comparator): To undergo the ELM procedure, the subject will sit comfortably in an exam chair.
  The Headset and Eye Pads will be adjusted to fit comfortably over gently closed eyelids. The subject will rest their head back. The ELM will be turned on, and will be active for 15 minutes wherein patients will feel a warming sensation to their eyes and a gentle vibration. The ELM is then removed.
  Interventions: Device: ELM
- Daily ELM Treatment (Active Comparator): To undergo the ELM procedure, the subject will sit comfortably in an exam chair.
  The Headset and Eye Pads will be adjusted to fit comfortably over gently closed eyelids. The subject will rest their head back. The ELM will be turned on, and will be active for 15 minutes wherein patients will feel a warming sensation to their eyes and a gentle vibration. The ELM is then removed. Subject will take personalized ELM home and use it as directed on a daily basis
  Interventions: Device: ELM

INTERVENTIONS:
Device: ELM — Treatment of dry eye with ELM device

SUMMARY:
The goal of this clinical trial is to evaluate the Eye Lipid Mobilizer (ELM) for the treatment of evaporative dry eye disease associated with meibomian gland dysfunction. The main questions aim to confirm that 1) the ELM can meet its intended use by validated patient reporting outcomes and 2) to confirm that the ELM device can be used safely by different users within a clinical environment as determined by review of any adverse events related to the use of the device.

DETAILED DESCRIPTION:
The purpose of the clinical study is to evaluate the Eye Lipid Mobilizer for the treatment of evaporative Dry Eye Disease associated with Meibomian Gland Dysfunction. The objective of the study is to confirm that the Eye Lipid Mobilizer (ELM) can meet its intended use by validated patient reporting outcomes.

The secondary objective is the ELM device can be used safety with no adverse events. The Eye Lipid Mobilizer (ELM) System is intended for the application of localized heat and vibration therapy in adult patients with chronic cystic conditions of the eyelids, including meibomian gland dysfunction (MGD), also known as evaporative dry eye or lipid deficiency dry eye.

ELIGIBILITY:
Inclusion Criteria:

* At least 21 years old
* Confirmed evaporative dry eye disease

Exclusion Criteria:

* Ocular surgery, trauma, herpes infections
* Unwillingness to comply with study protocol
* Pregnant or nursing women
* Any subject that cannot wear an eye mask
* Participation in another ophthalmic clinical trial within past 30 days

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Procedure-related adverse events | one week, four weeks
  Incidence of procedure-related adverse events will be assessed
Device-related adverse events | one week, four weeks
  Incidence of device-related adverse events will be assessed

SECONDARY OUTCOMES:
SPEED II Questionnaire for Dry Eye | one week, four weeks
  Change in outcomes for SPEED II Questionnaire for Dry Eye compared to baseline
Slip Lamp Evaluation | one week, four weeks
  Change of appearance of cornea under slit lamp evaluation compared to baseline
Meibomian Gland Imaging | one week, four weeks
  Change in meibomian gland under imaging compared to baseline
Lipid Layer Thickness | one week, four weeks
  Change in thickness of lipid layer compared to baseline
Tear Break Up Time | one week, four weeks
  Change in tear break up time compared to baseline
Corneal Fluorescein Staining | one week, four weeks
  Change in appearance of fluorescein staining compared to baseline

OTHER OUTCOMES:
Human Factors and Usability Evaluation | one week, four weeks
  Patients will participate in an Acceptance VAS Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: CEO, Study Director — Eyedetec
Locations (1):
- EYEcenter Optometric, Citrus Heights, California, United States

IPD SHARING:
Plan to Share IPD: No
will not be publishing in ICMJE journals

REFERENCES:
- [Result] Semeraro F, Forbice E, Braga O, Bova A, Di Salvatore A, Azzolini C. Evaluation of the efficacy of 50% autologous serum eye drops in different ocular surface pathologies. Biomed Res Int. 2014;2014:826970. doi: 10.1155/2014/826970. Epub 2014 Jul 22. PMID 25136628
- [Result] Finis D, Pischel N, Konig C, Hayajneh J, Borrelli M, Schrader S, Geerling G. [Comparison of the OSDI and SPEED questionnaires for the evaluation of dry eye disease in clinical routine]. Ophthalmologe. 2014 Nov;111(11):1050-6. doi: 10.1007/s00347-014-3042-z. German. PMID 25030896
- [Result] Savini G, Prabhawasat P, Kojima T, Grueterich M, Espana E, Goto E. The challenge of dry eye diagnosis. Clin Ophthalmol. 2008 Mar;2(1):31-55. doi: 10.2147/opth.s1496. PMID 19668387